CLINICAL TRIAL: NCT05768932
Title: A Phase 1 Study of BAL0891 as Monotherapy and in Combination With Chemotherapy or Tislelizumab in Patients With Advanced Solid Tumors or Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: BAL0891 in Patients With Advanced Solid Tumors or Relapsed or Refractory Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: SillaJen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TTK-CS-101
Record Dates: First submitted 2023-01-29; First posted 2023-03-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Tumor; TNBC - Triple-Negative Breast Cancer; Gastric Cancer; Leukemia Acute Myeloid Leukemia (AML)
Keywords: carcinoma; paclitaxel; BAL0891; tislelizumab
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Stomach Neoplasms; Leukemia, Myeloid, Acute; Carcinoma | interventions — tislelizumab; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part 1: Substudy 1, Dose-escalation substudy of BAL0891 monotherapy (Experimental): Increasing doses of BAL0891 will be administered IV on D1 and D8 Q3W (Regimen A). BAL0891 will be investigated in a dose range of 5-480 mg with Regimen A. Optionally, and based on cumulative safety, PK, and PD data, BAL0891 may be administered on D1 Q3W (Regimen B), D1 and D15 Q4W (Regimen C), or on D1, D8, and D15 Q4W (Regimen D).
  Interventions: Drug: BAL0891
- Part 1: Substudy 2, Dose-escalation substudy of BAL0891 in combination with tislelizumab (Experimental): Increasing doses of BAL0891 will be administrated IV on D1 and D15 with tislelizumab administration on D8 Q3W. The starting dose of BAL0891 for combination will be at approximately 50% of the BAL0891 monotherapy MTD determined in Substudy 1 and tislelizumab dose will be 200mg IV.
  Interventions: Drug: BAL0891; Combination Product: Tislelizumab
- Part 1: Substudy 3, Dose-escalation substudy of BAL0891 in combination with paclitaxel (Experimental): Paclitaxel will be dosed at 70 mg/m2 on D1, D8, and D15 Q4W, with an option to use 80 mg/m2 (either instead of, or after exploring, 70 mg/m2) if the cumulative data collected at that time support a higher dose of paclitaxel.
  Interventions: Drug: BAL0891; Combination Product: Paclitaxel
- Part 2 : Dose expansion, cohorts 1 TNBC (BAL0891 monotherapy) (Experimental): BAL0891 will be administered intravenously on D1 and D8, Q3W for cohorts 1. The investigation will focus on the RP2D determined during the dose escalation phase of the study. Specifically, cohorts 1 will utilize the RP2D established in substudy 1 of the dose escalation phase.
  Interventions: Drug: BAL0891
- Part 2 : Dose expansion, cohorts 2 GC (BAL0891 monotherapy) (Experimental): BAL0891 will be administered intravenously on D1 and D8, Q3W for cohorts 2. The investigation will focus on the RP2D determined during the dose escalation phase of the study. Specifically, cohorts 2 will utilize the RP2D established in substudy 1 of the dose escalation phase.
  Interventions: Drug: BAL0891
- Part 2 : Dose expansion, cohorts 3 TNBC (BAL0891 + Paclitaxel) (Experimental): BAL0891 will be administered intravenously on D1 and D15, Q4W for cohorts 3 . The investigation will focus on the RP2D determined during the dose escalation phase of the study. Specifically, cohorts 3 will utilize the RP2D established in substudy 3 of the dose escalation phase.
  Interventions: Drug: BAL0891; Combination Product: Paclitaxel
- Part 2 : Dose expansion, cohorts 4 GC (BAL0891 + Paclitaxel) (Experimental): BAL0891 will be administered intravenously on D1 and D15, Q4W for cohorts 4. The investigation will focus on the RP2D determined during the dose escalation phase of the study. Specifically, cohorts 4 will utilize the RP2D established in substudy 3 of the dose escalation phase.
  Interventions: Drug: BAL0891; Combination Product: Paclitaxel
- Part 1: Substudy 4, Dose-escalation substudy of BAL0891 monotherapy in r/r AML (Experimental): BAL0891 will be administered intravenously on Day 1 and Day 8 every three weeks (Regimen A). Dose exploration will proceed until the highest planned dose level (DL) is determined to be safe and tolerable, or the MTD/RP2D is identified.
  Interventions: Drug: BAL0891

INTERVENTIONS:
Drug: BAL0891 — BAL0891 is a dual inhibitor of threonine tyrosine kinase (TTK) and polo-like kinase 1 (PLK1)
  Other Names: TTK-CS-101
Combination Product: Tislelizumab — Tislelizumab a humanized IgG4 anti-PD-1 monoclonal antibody
  Arms: Part 1: Substudy 2, Dose-escalation substudy of BAL0891 in combination with tislelizumab
Combination Product: Paclitaxel — Paclitaxel is a natural product with antitumor activity
  Other Names: Taxol
  Arms: Part 1: Substudy 3, Dose-escalation substudy of BAL0891 in combination with paclitaxel; Part 2 : Dose expansion, cohorts 3 TNBC (BAL0891 + Paclitaxel); Part 2 : Dose expansion, cohorts 4 GC (BAL0891 + Paclitaxel)

SUMMARY:
This study is a multiple cohort, multicenter, open-label Phase 1 study with dose-escalation substudies investigating intravenous (IV) BAL0891 as monotherapy, and in combination with tislelizumab or paclitaxel, to determine the safety and tolerability of increasing doses of BAL0891 in patients with advanced solid tumors or relapsed or refractory acute myeloid leukemia. An adaptive model-based design will be used to guide the dose escalation. Subject assignment to Substudy 1, 2, 3 and 4 will be finalized following approval from the investigator and sponsor.

The dose-expansion stage will be conducted with the RP2D to further evaluate the preliminary anti-tumor activity, safety, and tolerability in metastatic TNBC and GC.

DETAILED DESCRIPTION:
Substudy 1 (monotherapy dose-escalation cohorts) This study will be initiated with enrollment into Substudy 1 and will estimate the safety, tolerability, PK, and PD of increasing doses of BAL0891 in patients with advanced solid tumors. The starting dose will be 5 mg based on the GLP (Good Laboratory Practice) toxicology studies. Dose escalation will comprise a dose range from a dose of 5 mg up to a maximum absolute dose of 480 mg, with eight nominal dose levels (DLs) of 5 / 10 / 20 / 40 / 80 / 160 / 320 / 480 mg. Intra-patient dose escalations are only allowed for patients enrolled in single-patient DL Cohorts 1.1, 1.2, and 1.3. From DL Cohort 1.4 onwards, the projected maximum dose-escalation factor will be two-fold; if the DL cohort investigates an increased dose, dosing of the patients within the cohort must be separated by at least 7 days. For cohorts in which doses are not increased (including backfill enrollment), patients may be enrolled concurrently.

BAL0891 will be administered intravenously (IV) on Day (D) 1 and D8 every 3 weeks (Q3W); for the schedule of assessments of Regimen A. Alternative 21-day or 28-day dosing regimens may be investigated; for the schedule of assessments of Regimens B-D.

Substudies 2 and 3 (dose-escalation cohorts for combination regimens) Enrollment into Substudies 2 and 3 may commence as early as first signs of expected target toxicity and/or efficacy with Regimen A (or an alternative monotherapy regimen) have been observed, or alternatively, once the MTD of BAL0891 monotherapy has been assessed. Patients enrolled into Substudies 2 and 3 will be treated with increasing doses of BAL0891 in combination with tislelizumab or paclitaxel, respectively, and dose escalation of both BAL0891 and tislelizumab/paclitaxel if required will use the same cumulative BLRM-EWOC model as Substudy 1. The starting dose of BAL0891 in combination with tislelizumab or paclitaxel will be a safe DL determined in Substudy 1 but not higher than approximately half the MTD. Backfill enrollment of up to a total of 30 additional patients for both substudies (who may be enrolled concurrently) may be used to better estimate the RP2D for each combination if required.

Substudy 4 (dose escalation cohort for monotherapy in r/r AML) Substudy 4 will evaluate BAL0891 monotherapy in patients with relapsed/refractory AML (r/r AML) using the same BLRM-EWOC model and study design described for Substudy 1. BAL0891 will be administered intravenously on Day 1 and Day 8 every three weeks (Regimen A; see Table 13 for schedule of assessments). Dose exploration will proceed until the highest planned dose level (DL) is determined to be safe and tolerable, or the MTD/RP2D is identified.

Each DL cohort will enroll three patients, with DLT observation required before advancing to the next DL. From DL2 onward, the projected maximum dose-escalation factor will be two-fold, with concurrent enrollment allowed for cohorts without dose increases. Backfill enrollment may be conducted to refine the RP2D and further characterize safety, efficacy and PD.

Part 2 : Dose expansion The commencement of the dose expansion stage will follow the determination of the RP2D achieved during the dose-escalation phase. This stage will consist of four cohorts, each comprising 24 patients who have previously undergone at least one systemic regimen for advanced or metastatic disease. Specifically, two cohorts will be allocated for TNBC, investigating BAL0891 both as a monotherapy and in combination with Paclitaxel. Additionally, two cohorts will be designated for GC, investigating the outcomes of BAL0891 as a monotherapy and in combination with Paclitaxel.

ELIGIBILITY:
1.1. Inclusion criteria: Substudy 1, 2, 3 and Dose expansion Each patient must meet all the following inclusion criteria.

1. Informed consent signed by the patient prior to any study-related procedure indicating that they understand the purpose of, and procedures required for, the study, and are willing to participate in the study.
2. Male or female aged ≥18 years (or ≥ 19 years according to local regulatory guidelines) at the time of screening.
3. Patients with incurable advanced/metastatic solid tumor disease refractory to or intolerant of existing therapy known to provide clinical benefit for their condition.

   Note: Patients with non-CNS tumors participating during dose escalation may have inactive CNS metastasis, defined as 4 weeks after either brain metastasis resection or radiation, and a) all residual neurological symptoms resolved to grade ≤ 2; b) on stable doses of dexamethasone, if applicable; and c) follow-up imaging shows no new lesions appearing.
4. Patients enrolled in Dose Expansion only

   • TNBC cohorts i. Must have histologically confirmed breast adenocarcinoma that is unresectable, loco-regional, or metastatic.

   ii. Must have source data documented pathologically confirmed triple negative breast cancer, defined as both of the following.
   1. Estrogen receptor (ER) and progesterone receptor (PgR) negative: <1% of tumor cell nuclei are immunoreactive in the presence of evidence that the sample can express ER or PgR (positive intrinsic controls)
   2. Human epidermal growth factor receptor 2 (HER2) negative as per American Society of Clinical Oncology/College of American Pathologists guidelines

      * IHC 0 or 1 fluorescence in situ hybridization (FISH) negative (or equivalent negative test)
      * Patients with IHC 2 must have a negative by FISH (or equivalent negative test) iii. Patients with a history of different breast cancer phenotypes (i.e., ER/PgR/HER2 Positive) must obtain pathological confirmation of triple-negative disease in at least one of the current sites of metastasis.

   iv. Must have progression on or after therapy containing anthracycline and/or a taxane. Subjects must have received anthracycline and/or a taxane based regimen or other chemotherapy / targeted therapy regimen if anthracycline or taxane was contraindicated or another available approved targeted agent was contraindicated. At time of enrolment, patients must have progressed on, be intolerant of, or be ineligible for, all available standard of care therapies with proven benefit.

   • GC cohort i. Must have a histologically or cytologically confirmed diagnosis of gastric or gastroesophageal junction adenocarcinoma.

   ii. Must have progression on or after therapy containing platinum/fluoropyrimidine. Subjects must have received platinum-based chemotherapy or other chemotherapy regimen if platinum-based chemotherapy was contraindicated or another available approved targeted agent unless the targeted agent was contraindicated. At time of enrolment, patients must have progressed on, be intolerant of, or be ineligible for, all available standard of care therapies with proven benefit.

   iii. Documentation of HER2/neu status. Patients who are HER2/neu-positive must be treated with a HER2/neu inhibitor, and subjects should have progressed on or be intolerant to the targeted therapy or subjects must have received other chemotherapy regimen if HER2/neu inhibitor was contraindicated or another available approved targeted agent unless the targeted agent was contraindicated. At time of enrolment, patients must have progressed on, be intolerant of, or be ineligible for, all available standard of care therapies with proven benefit.

   iv. Subjects must/should have received no more than 3 lines of prior therapy for the advanced disease (if a subject progressed within 6 months of completing adjuvant therapy, this would count as a prior line of therapy).
5. For patients enrolled in Substudy 3 or cohort 3 and 4, if a taxane (i.e., paclitaxel or docetaxel) was administered as part of the previous regimen, PD must have occurred > 12 months from the end of the previous treatment. (Patients who received a taxane in previous treatments without reaching PD may enroll without the 12-month waiting period.)
6. Patients enrolled in Dose Expansion only, patient must have undergone a minimum of 1 prior systemic regimen for advanced or metastatic disease. (Korea only, patients must have received the second line standard of care treatment as per the regulations of the respective country. Patients who are unsuitable to receive the standard of care second line treatment will be eligible for enrollment)
7. Eastern Cooperative Oncology Group performance status (ECOG PS) 0or-1
8. For patients enrolled from DL1.4 of Substudy 1 onwards and for all patients in Substudies 2 and 3 and all four dose expansion cohorts, measurable tumor disease per Response Evaluation Criteria in Solid Tumors 1.1 criteria (RECIST 1.1), i.e., a minimum of one target lesion.
9. Adequate organ functions as indicated by the following Screening visit local laboratory values:

   1. Hemoglobin ≥ 9 g/dL (criterion must be met without erythropoietin dependency and without packed red blood cell transfusion within the last 4 weeks)
   2. ANC ≥ 2.0 × 109/L; criterion must be met without growth factor (e.g., G-CSF, GM CSF, etc.) administration within the last 2 weeks
   3. Platelets ≥ 100 × 109/L
   4. Total bilirubin ≤ 1.5 × ULN
   5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) baseline levels ≤ 1.5 × ULN, with the option for AST/ALT ≤ 3.0 × ULN, or ≤ 5.0 × ULN for patients with liver metastasis, upon accumulating evidence for the absence of liver toxicity in biologically active DLs
   6. Albumin ≥ 2.8 g/dL
   7. CLCR ≥ 50 mL/min (as calculated by the Cockcroft-Gault formula), or eGFR ≥ 50 mL/min/1.73 m² (MDRD equation or CKD-EPI equation)
   8. For women of childbearing potential, negative serum human chorionic gonadotropin (hCG)
10. Men/women of child-producing/bearing potential must agree to: avoid impregnating a partner or becoming pregnant, respectively, during the study, and for at least 6 months after the last dose of either investigational drug, and comply with the contraception requirements.

1.2. Inclusion criteria: Substudy 4 Each patient must meet all the following inclusion criteria.

1. Informed consent signed by the patient prior to any study-related procedure indicating that they understand the purpose of, and procedures required for, the study, and are willing to participate in the study.
2. Male or female aged ≥18 years (or ≥ 19 years according to local regulatory guidelines) at the time of screening.
3. Eastern Cooperative Oncology Group performance status (ECOG PS) 0-2.
4. Estimated life expectancy of at least 8 weeks
5. AML either de novo or secondary as any subtype diagnosed according to the WHO 2022 classification system [except acute promyelocytic leukemia (APL)] who either:

   Relapse/refractory (R/R) acute myeloid leukemia (AML) defined as those who have also failed or are not appropriate for any approved standard-of-care (SOC) therapies, or hematopoietic stem cell transplant (HSCT) with reappearance of ≥ 5% blasts in the bone marrow.
6. Relapsed AML is defined as having 5% or more leukemic blasts in the bone marrow, reappearance of leukemic blasts in peripheral blood (in at least two peripheral blood samples taken at least one week apart), or the development of new extramedullary disease.
7. WBC, peripheral blood leukocyte count≤ 25,000/µL and blast count ≤ 25,000/µL prior to initiation of therapy

   1. Hydroxyurea is allowed during screening and prior to day 1 of study treatment to keep the blast count ≤25,000/µL; hydroxyurea is to be ceased 24 hours prior to study therapy.
   2. Hydroxyurea may be used for up to 28 days in the initial treatment cycle if needed, to keep the white blood cell (WBC) count ≤25,000/µL. However, no other anti-leukemic treatments, apart from the study drug, are allowed during this period.
   3. Leukapheresis is allowed to maintain blast count ≤25,000/µL
8. Adequate organ functions as indicated by the following Screening visit local laboratory values:

   1. CLCR ≥ 60 mL/min (as calculated by the Cockcroft-Gault formula), or eGFR ≥ 60 mL/min/1.73 m² (MDRD equation or CKD-EPI equation)
   2. Total bilirubin ≤ 1.5 × ULN (unless considered due to leukemic organ involvement), or, Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
   3. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) baseline levels ≤ 3.0 × ULN
   4. Albumin ≥ 2.5 g/dL
   5. International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
   6. Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
9. Men/women of child-producing/bearing potential must agree to: avoid impregnating a partner or becoming pregnant, respectively, during the study, and for at least 6 months after the last dose of either investigational drug, and comply with the contraception requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2022-12-14 (Actual); Primary Completion 2026-12-24 (Estimated); Study Completion 2026-12-24 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants With Adverse Events as a Measure of Safety and Tolerability | After first dose, up to 2 years
  Safety is collected through summaries of AE(Adverse Event)s, safety laboratory evaluations, PK evaluations, physical examinations, vital signs, and ECGs using CTCAE v5.0.
Part 1: Number of Participants With the DLT (Dose-limiting toxicity)s as a Measure of maximum tolerated dose (MTD) and/or the recommended Phase 2 dose (RP2D) | After first dose and within 7 days of End of Treatment, up to 2 years
  DLTs are collected through BLRM-EWOC.
Part 2: Overall response rate (ORR) for all subjects | Every 3 months (±14 days) after first dose, up to 2 years
  The proportion of patients with confirmed complete response (CR) or partial response (PR) by RECIST 1.1/iRECIST (substudy 2 only) during the dose expansion phase.

SECONDARY OUTCOMES:
Part 1: Pharmacokinetics (PK) parameters for all subjects | Within 7 days of End of Treatment, up to 2 years
  The area under the plasma concentration-time curve (AUC) by PK Sampling
Part 1: Absolute neutrophil count (ANC) for all subjects | Within 7 days of End of Treatment, up to 2 years
  Duration of neutropenia by PD Sampling
Part 1, 2: Overall response rate (ORR) for all subjects | Every 3 months (±14 days) after first dose, up to 2 years
  The proportion of patients with confirmed complete response (CR) or partial response (PR) by RECIST 1.1
Part 1, 2: Disease control rate (DCR) for all subjects | Within 7 days of End of Treatment, up to 2 years
  The proportion of patients with confirmed CR, PR or stable disease (SD) by RECIST 1.1
Part 1, 2: Progression-free survival (PFS) for all subjects | Within 7 days of End of Treatment, up to 2 years
  Measured from patient enrollment to disease progression date
Part 1, 2: Overall survival (OS) for all subjects | Within 7 days of End of Treatment, up to 2 years
  Measured from from patient enrollment to time of death
Part 2: Safety evaluations for all subjects | After first dose, up to 2 years
  Safety evaluations is focusing on key clinical evlauations such treatment-emergent adverse events (TEAE) using CTCAE v5.0.
Part 1: Efficacy Endpoints CR + CRh Rate (Substudy 4) | Up to 2 years
  Proportion of patients achieving Complete Remission (CR) or CR with partial hematologic recovery (CRh) per European LeukemiaNet (ELN) 2022 guidelines.
Part 1: Efficacy Endpoints Duration of Remission (DoR) (Substudy 4) | Up to 2 years
  Time from first documented CR/CRh until relapse or death.
Part 1: Efficacy Endpoints Transfusion Independence (TI) (Substudy 4) | Up to 2 years
  Proportion of patients achieving red blood cell (RBC) and platelet transfusion independence for ≥56 consecutive days.
Part 1: Efficacy Endpoints CR/CRh without Measurable Residual Disease (MRD) (Substudy 4) | Up to 2 years
  Proportion of patients achieving CR/CRh and MRD negativity.
Part 1: Efficacy Endpoints Composite Complete Remission (CRc) Rate (Substudy 4) | Up to 2 years
  Proportion of patients achieving CR, CRh, or CR with incomplete hematologic recovery (CRi).
Part 1: Efficacy Endpoints Overall Response Rate (ORR) (Substudy 4) | Up to 2 years
  Proportion of patients achieving CR, CRh, CRi, or Partial Remission (PR).
Part 1: Efficacy Endpoints Overall Survival (OS) (Substudy 4) | Up to 2 years
  Time from first dose of BAL0891 to death from any cause.
Part 1: Efficacy Endpoints Event-Free Survival (EFS) (Substudy 4) | Up to 2 years
  Time from first dose of BAL0891 to disease progression, relapse, or death.
Part 1: Efficacy Endpoints Time to Response (TTR) (Substudy 4) | Up to 2 years
  Time from first dose of BAL0891 to first documented response.
Part 1: QTcF Interval Analysis | From first dose to 30 days post last dose
  Analysis of QTcF interval data collected during BAL0891 monotherapy and the relationship between BAL0891 exposure and QTcF interval prolongation.

CONTACTS AND LOCATIONS:
Overall Officials: SillaJen Inc., Study Director — SillaJen, Inc.
Locations (12):
- United States (6):
  - Yale New Haven Hospital, New Haven, Connecticut
  - University of Miami Health System, Coral Gables, Florida
  - Montefiore Medical Center, The Bronx, New York
  - OHSU Knight Cancer Institute, Portland, Oregon
  - Mary Crowley Cancer Research, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- South Korea (6):
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Asan Medical Center, Seoul
  - Korean University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul

IPD SHARING:
Plan to Share IPD: No